CLINICAL TRIAL: NCT02916732
Title: Études Observationnelles Des conséquences de l'Infection à Virus Zika au Cours de la Grossesse Pendant l'épidémie Des départements français d'Amérique de l'année 2016
Brief Title: Zika Virus Infection's Pregnancy Consequences in French Department of America
Acronym: ZIKA-DFA-FE
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C16-08; 2016-A00399-42 (Other: France ANSM)
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2022-05

CONDITIONS: Incidence of ZIKV Infection on Fetus During the Pregnancy
Keywords: asymptomatics; microcephaly; abnormalities
MeSH Terms: conditions — Microcephaly; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — * bio-bank of serum from all pregnant women.
  * bio-bank of maternal blood and infant cord blood
  * bio-bank of maternal blood and fetal tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Module 1: Identification and monitoring of pregnant women who develop clinical signs of acute infection due to ZIKV (standard monitoring report)
- Module 2: Monitoring of pregnant women with a suspected embryofetopathy (standard monitoring report)
- Module 3: Trimester biological collection of all pregnant women during the outbreak of Zika (standard monitoring report)
- Module 4: Biological collection of maternal blood and cord blood collected during the delivery
- Module 5: Biological collection of maternal blood and fetal tissues of pregnant women whose pregnancies started during the outbreak of Zika , ends in an spontaneous abortion, Induced abortion or intrauterine fetal demise

SUMMARY:
The Zika (ZIKV) epidemic has spread into the three French Overseas Departments in the Caribbean (DFAs). It is therefore urgent to set up tools to collect clinical and paraclinical data for the evaluation of potential complications due to having ZIKV infection during pregnancy. This study is meant to collect, within usual care practices, clinical and paraclinical information which will allow the precise description of the consequences of ZIKV infection occurring during pregnancy.

DETAILED DESCRIPTION:
This is a prospective observational, non-interventional study that has been integrated into the usual standard of care practices. All information and biological samples collected during the course of this project will be done through the new medical standard of care which has been put in place during the ZIKV epidemic in the DFAs; this new standard of care is a result of existing recommendations from medical professionals and/or public health authorities. Outside of these recommendations, no invasive procedure will be done simply to satisfy an objective of this study.

ELIGIBILITY:
M1:

Inclusion Criteria:

* On-going pregnancy regardless the presumed date of birth
* Clinical signs suggestive of ZIKV infection
* Whatever the RT-PCR analysis

Exclusion Criteria:

* Minor
* No consent

M2:

Inclusion Criteria:

* Head circumference < 5th percentile
* Other brain morphological abnormality
* Hydramnios
* Intrauterine growth restriction (IUGR)

Exclusion Criteria:

* Minor
* No consent

M3:

Inclusion Criteria:

* Pregnant woman during epidemic period of ZIKV

Exclusion Criteria:

* Minor
* Opposition

M4:

Inclusion Criteria:

* Delivery during epidemic period of ZIKV

Exclusion Criteria:

* Minor
* No consent

M5:

Inclusion Criteria:

* Spontaneous abortion or fetal death in utero during epidemic period of ZIKV

Exclusion Criteria:

* Minor
* No consent

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of this study is women who have been pregnant during the 2016 ZIKV Epidemic in the DFAs. Five study arms (hereafter called 'modules') have been defined with various inclusion criteria for each module.
  M1: Pregnant women with clinical signs of acute ZIKV infection
  Module 2: Pregnant women for which an abnormality has been detected in the fetus.
  Module 3: Bio-bank of serum, collected once per trimester, from all pregnant women.
  Module 4: Bio-bank of maternal blood and infant cord blood, taken the day of birth in all mothers and their babies in the 3 DFAs.
  Module 5: Bio-bank of maternal blood and fetal tissues from women in whom the pregnancy was terminated due to miscarriage, abortion on medical grounds, or a fetal death in-utero.
Sampling Method: Non-Probability Sample
Enrollment: 26980 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Incidence of ZIKV infection during pregnancy | 12 months

SECONDARY OUTCOMES:
Incidence of microcephaly and other fetal abnormalities | 12 month

OTHER OUTCOMES:
Analysis of risk factor for the occurence of congenital abnormalities | 12 month

CONTACTS AND LOCATIONS:
Locations (4):
- French Guiana (2):
  - CH Andrée Rosemon (CHAR), Cayenne
  - CH de l'Ouest Guyanais Franck Joly (CHOG), Saint-Laurent-du-Maroni
- CHU de Pointe à Pitre/Les Abymes, Pointe-à-Pitre, Guadeloupe
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Funk AL, Hoen B, Vingdassalom I, Ryan C, Kadhel P, Schepers K, Gaete S, Tressieres B, Fontanet A. Reassessment of the risk of birth defects due to Zika virus in Guadeloupe, 2016. PLoS Negl Trop Dis. 2021 Mar 3;15(3):e0009048. doi: 10.1371/journal.pntd.0009048. eCollection 2021 Mar. PMID 33657112
- [Result] Hoen B, Schaub B, Funk AL, Ardillon V, Boullard M, Cabie A, Callier C, Carles G, Cassadou S, Cesaire R, Douine M, Herrmann-Storck C, Kadhel P, Laouenan C, Madec Y, Monthieux A, Nacher M, Najioullah F, Rousset D, Ryan C, Schepers K, Stegmann-Planchard S, Tressieres B, Volumenie JL, Yassinguezo S, Janky E, Fontanet A. Pregnancy Outcomes after ZIKV Infection in French Territories in the Americas. N Engl J Med. 2018 Mar 15;378(11):985-994. doi: 10.1056/NEJMoa1709481. PMID 29539287